CLINICAL TRIAL: NCT00668291
Title: Assessment of the Clinical Symptoms of the Primary Pigmented Nodular Adrenocortical Disease (PPNAD) and the CARNEY Complex (CNC).
Brief Title: Primary Pigmented Nodular Adrenocortical Disease (PPNAD) and the CARNEY Complex (CNC)
Acronym: EVACARNEY
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: P060251
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Primary; Complex; Pigmented Nodular Adrenocortical Disease, Primary, 1; Periorificial Lentiginosis; Cardiac Myxoma
Keywords: Endocrinology, CARNEY Complex,; primary pigmented nodular adrenocortical disease (PPNAD),; PRKAR1A
MeSH Terms: conditions — Pigmented Nodular Adrenocortical Disease, Primary, 1; Carney Complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 2 tubes EDTA 5 mL each (DNA) and 2 tubes heparine 5 mL each (cellular biology)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CNC: Primary pigmented nodular adrenocortical disease (PPNAD) and the Carney complex (CNC)
- MC-L: cardiac myxoma or isolated lentiginosis

SUMMARY:
Cohort CNC-PPNAD will be investigated with clinical, genetic, biological and imaging work-up every year during 3 years. Cohort L-MC will be investigated clinically at inclusion and a PERKAR1A genotype will be performed.

DETAILED DESCRIPTION:
The primary aim is to assess the clinical manifestations of the CARNEY Complex (CNC) and/or the primary pigmented nodular adrenocortical disease (PPNAD) in patients with CNC, isolated PPNAD or carriers of PRKAR1A and PPNAD1 (PDE11A4) germline mutation (Cohort CNC-PPNAD). In this cohort genotype/phenotype correlation will be studied. A second aim is to determine the frequency of PRKAR1A germline mutation in patients with isolated cardiac myxoma or isolated lentiginosis (Cohort L-MC).

ELIGIBILITY:
Inclusion Criteria:

CNC group :

* patient with the CARNEY complex (CNC) or the primary pigmented nodular adrenocortical disease (PPNAD) or a germinal mutation of the gene of CARNEY Complex or PPNAD.
* No age criteria
* Inform consent of the patient or the parental authority collected
* Realization of a preliminary medical examination
* Affiliated with a social security system ( profit or having right)

MC-L group :

* Patient with periorificial lentiginosis or cardiac myxoma
* or previous history of periorificial lentiginosis or cardiac myxoma
* age > or = 18 years old
* Realization of a preliminary medical examination
* Affiliated with a social security system ( profit or having right)

Exclusion criteria :

CNC group and MC-L group:

* refusal or incapacity to take part in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consultations
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2008-01; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To assess the clinical manifestations of the CARNEY Complex (CNC) and/or the primary pigmented nodular adrenocortical disease (PPNAD) | 6 months

SECONDARY OUTCOMES:
Genotype/phenotype correlation. To determine the frequency of PRKAR1A germline mutation in patients with isolated cardiac myxoma or isolated lentiginosis. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Bertherat, MD PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

REFERENCES:
- [Result] Espiard S, Vantyghem MC, Assie G, Cardot-Bauters C, Raverot G, Brucker-Davis F, Archambeaud-Mouveroux F, Lefebvre H, Nunes ML, Tabarin A, Lienhardt A, Chabre O, Houang M, Bottineau M, Stroer S, Groussin L, Guignat L, Cabanes L, Feydy A, Bonnet F, North MO, Dupin N, Grabar S, Duboc D, Bertherat J. Frequency and Incidence of Carney Complex Manifestations: A Prospective Multicenter Study With a Three-Year Follow-Up. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgaa002. doi: 10.1210/clinem/dgaa002. PMID 31912137
- [Result] Bertherat J. Carney complex (CNC). Orphanet J Rare Dis. 2006 Jun 6;1:21. doi: 10.1186/1750-1172-1-21. PMID 16756677
- [Result] Kirschner LS, Carney JA, Pack SD, Taymans SE, Giatzakis C, Cho YS, Cho-Chung YS, Stratakis CA. Mutations of the gene encoding the protein kinase A type I-alpha regulatory subunit in patients with the Carney complex. Nat Genet. 2000 Sep;26(1):89-92. doi: 10.1038/79238. PMID 10973256
- [Result] Carney JA, Gordon H, Carpenter PC, Shenoy BV, Go VL. The complex of myxomas, spotty pigmentation, and endocrine overactivity. Medicine (Baltimore). 1985 Jul;64(4):270-83. doi: 10.1097/00005792-198507000-00007. PMID 4010501
- [Derived] Vaduva P, Violon F, Jouinot A, Bouys L, Espiard S, Bonnet-Serrano F, North MO, Cardot-Bauters C, Raverot G, Hieronimus S, Lefebvre H, Nunes ML, Tabarin A, Groussin L, Assie G, Sibony M, Vantyghem MC, Pasmant E, Bertherat J. Carney complex predisposes to breast cancer: prospective study of 50 women. Eur J Endocrinol. 2024 Feb 1;190(2):121-129. doi: 10.1093/ejendo/lvae010. PMID 38252880